CLINICAL TRIAL: NCT03641430
Title: The Effects of Over-the-Counter Products on the Skin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study design will need to be changed completely becasue of the change of research interest. We have decided to withdraw the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00180361
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Skin Health
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care with Over-the-Counter (OCT) product (Experimental): Participants will apply over-the-counter product for a certain period with or without light challenge
  Interventions: Other: Supportive care with OCT product

INTERVENTIONS:
Other: Supportive care with OCT product — Participants will apply over-the-counter product for a certain period with or without light challenge. We will perform clinical assessments of the skin associated with product application as well as assess these changes with and without light challenge. Skin biopsies will be obtained following standard medical practice and will be used to analyze skin markers related to photoaging, pigmentation, oxidative stress, and other dermatologic conditions.

SUMMARY:
The primary purpose of this study is to investigate the safety and tolerability of commonly used over-the-counter products and the effects of the products on skin health.

DETAILED DESCRIPTION:
Participant will apply commonly used skin product on skin for a period of time with or without light challenge. The investigators will perform clinical assessments of the skin associated with product application as well as assess these changes with and without light challenge. Skin biopsies will be obtained following standard medical practice and will be used to analyze skin markers related to photoaging, pigmentation, oxidative stress, and other dermatologic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 years old with healthy skin;
* Participant must be willing and comply with the requirements of the protocol;
* Participant must have the ability to understand and communicate with the investigator;
* Participant must provide informed consent.

Exclusion Criteria:

* Subjects who are unable to provide informed consent;
* Subject with significant medical history or current skin diseases that the investigator feels is not safe for study participation;
* Subjects who self-report that they are pregnant or nursing;
* Subjects who do not speak English or have difficulty hearing or are otherwise impaired for providing informed consent and communicating with the investigator;
* Subjects with known bleeding disorders or diathesis;
* Subjects with a history of keloids or excessive scarring;
* Subjects with known allergy to lidocaine, epinephrine, or any of the tested products;
* Subjects who foresee intensive UV exposure during the study (e.g. sunbathing, tanning beds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Photoaging | 1 year
  This will be assessed using the Griffiths Photoaging Photonumeric scale with range from 1 to 10 with increasing numbers representing advanced photoaging

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chien, Principal Investigator — Johns Hopkins University
Locations (1):
- Cutaneous Translational Research Program, Department of Dermatology, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor EC, Watson RE, Sherratt MJ. Molecular aspects of skin ageing. Maturitas. 2011 Jul;69(3):249-56. doi: 10.1016/j.maturitas.2011.04.011. Epub 2011 May 25. PMID 21612880